## **Overview of Study Documents**

A Multicenter, Adaptive, Randomized,
Blinded Controlled Trial of the Safety and
Efficacy of Investigational Therapeutics for
Hospitalized Patients with Acute
Respiratory Distress Syndrome Associated
with COVID-19

**05 August 2025** 

NCT06729593

(Master protocol: NCT04843761)

## ACTIV-3b: Therapeutics for Severely Ill Inpatients With COVID-19 (TESICO) trial.

## **Overview of Trial Documents**

Master protocol: NCT04843761 Aviptadil Substudy (H1): NCT06729606 Remdesivir Substudy (H2): NCT06729593

| Document | Document Date | Description |
|---|---|---|
| Study Protocol: Master | March 8, 2022 | The master protocol document for TESICO/ACTIV-3b. |
| | | This document should be used together with the agent specific appendices (H1 and H2) to understand the data collection for the Aviptadil and Remdesvir substudies. |
| Study Protocol:<br>Aviptadil (H1) | March 8, 2022 | Appendix H1 to the TESICO master protocol document. Provides additional agent-specific information for the Aviptadil component of the trial. |
| Study Protocol:<br>Remdesivir (H2) | April 1, 2021 | Appendix H2 to the TESICO master protocol document. Provides additional agent-specific information for the Remdesivir component of the trial and a description of the 4 randomization strata used for enrollment into both agents. |
| Statistical Analysis<br>Plan: Main | August 5, 2021 | This document applies for both the Aviptadil and Remdesivir substudies. |
| Statistical Analysis<br>Plan: Addendum | May 1, 2022 | This document applies to the Aviptadil substudy. |
| Informed Consent | March 8, 2022 | This document applies for both the Aviptadil and Remdesivir substudies. |